CLINICAL TRIAL: NCT07287293
Title: Comparison of Endotracheal Tube Suctioning Versus No Suctioning During Emergence From General Anesthesia With Endotracheal Intubation: A Randomized, Single-Blind Study
Brief Title: Endotracheal Tube Suctioning Versus No Suctioning During Emergence From General Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Suction
Record Dates: First submitted 2025-11-15; First posted 2025-12-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hypoxia; Airway Obstruction, Postoperative; Sore Throat; Cough, Postoperative
Keywords: Airway Management; Suctioning; Emergence from Anesthesia; Hypoxia; Endotracheal Intubation; Postoperative Complications
MeSH Terms: conditions — Hypoxia; Airway Obstruction; Pharyngitis; Cough; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Interventions
  Routine Suctioning Group (SUC):
  Participants received both endotracheal suctioning and oropharyngeal suctioning immediately prior to extubation, performed using standard suction pressure and technique.
  No Suctioning Group (NON-SUC):
  Participants received oropharyngeal suctioning only. No suction catheter was inserted into the trachea prior to extubation.
  If the anesthesiologist identified copious airway secretions requiring clearance for patient safety, endotracheal suctioning was performed. These participants were subsequently excluded from the analysis as per the predefined protocol.
Who Masked: Outcomes Assessor
Masking Description: The anesthesiologist performing the intervention, the participants, and the investigators involved in intraoperative care and data collection were not masked because the suctioning procedures could not be concealed. The outcomes assessor, responsible for recording postoperative oxygen saturation, airway symptoms, and patient-reported outcomes, was blinded to the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Endotracheal Suctioning (SUC) (Active Comparator): Participants in this arm received routine endotracheal suctioning immediately prior to extubation, performed using standard suction pressure and technique. Oropharyngeal suctioning was also performed according to usual clinical practice.
  Interventions: Procedure: Routine Endotracheal Suctioning
- Omission of Endotracheal Suctioning (NON-SUC) (Experimental): Participants in this arm received oropharyngeal suctioning only prior to extubation. No suction catheter was inserted into the trachea. Standard anesthetic care and monitoring were provided as per routine practice.
  Interventions: Procedure: Omission of Endotracheal Suctioning

INTERVENTIONS:
Procedure: Routine Endotracheal Suctioning — Endotracheal suctioning performed immediately prior to extubation using standard suction pressure and technique. Oropharyngeal suctioning was also performed according to routine clinical practice.
  Other Names: SUC
  Arms: Routine Endotracheal Suctioning (SUC)
Procedure: Omission of Endotracheal Suctioning — Oropharyngeal suctioning only was performed prior to extubation. No suction catheter was inserted into the trachea.
  Other Names: NON-SUC
  Arms: Omission of Endotracheal Suctioning (NON-SUC)

SUMMARY:
The goal of this study is to determine whether omitting tracheal suctioning immediately prior to extubation is non-inferior to routine tracheal suctioning with respect to early postoperative oxygenation among adult surgical patients (aged 18-90 years, American Society of Anesthesiologists [ASA] physical status I-III) undergoing elective surgery under general anesthesia with endotracheal intubation.

The study addresses the following questions:

* Primary outcome (non-inferiority):
* Is the risk of postoperative desaturation (oxygen saturation [SpO₂] <92% within 60 minutes after extubation) in the no-suction group not worse than in the routine-suction group by more than 10 percentage points?
* Secondary outcomes (superiority):
* Does omitting tracheal suctioning reduce postoperative cough severity and sore throat?
* Does omitting tracheal suctioning avoid increasing extubation-related adverse events?

Participants will be randomly assigned (1:1) to one of two groups:

* Routine suctioning (SUC): Endotracheal suctioning plus oropharyngeal suctioning immediately before extubation
* No suctioning (NON-SUC): Oropharyngeal suctioning only, without endotracheal suctioning

All participants will receive standard anesthetic care and postoperative monitoring in the post-anesthesia care unit (PACU) for 60 minutes. Follow-up for airway symptoms and patient satisfaction will be conducted at 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-90 years with American Society of Anesthesiologists (ASA) physical status I-III.
* Scheduled for elective surgery under general anesthesia requiring endotracheal intubation.
* Planned tracheal extubation in the operating room at the end of surgery.

Exclusion Criteria:

* Inability to provide informed consent or the presence of a significant language barrier that prevents effective communication with the clinical team.
* Known diagnosis of obstructive sleep apnea (OSA), active pneumonia, or chronic pulmonary disease (e.g., chronic obstructive pulmonary disease, restrictive lung disease).
* Body mass index (BMI) >35 kg/m².
* Pregnancy or increased aspiration risk (e.g., full stomach).
* Scheduled for maxillofacial, head and neck, or airway surgery.
* Anticipated surgical duration >3.5 hours.
* Anticipated difficult airway, defined as the presence of ≥2 predictors of difficult mask ventilation (DMV) based on Langeron et al., or a documented history of difficult intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative desaturation after extubation | First 60 minutes after extubation
  Proportion of participants who develop desaturation, defined as peripheral oxygen saturation (SpO₂) <92% at any time within the first 60 minutes after extubation.

SECONDARY OUTCOMES:
Incidence and severity of postoperative coughing | First 60 minutes after extubation
  Incidence and severity of postoperative coughing within the first 60 minutes after extubation, assessed using the modified Minogue scale. Severity is recorded as the highest coughing score observed during the assessment period.
Severity of sore throat during swallowing | First 60 minutes after extubation
  Severity of sore throat during swallowing within the first 60 minutes after extubation, assessed using a 0-10 numerical rating scale (NRS). The outcome is recorded as the highest score reported during the assessment period.
Requirement and level of oxygen therapy | First 60 minutes after extubation
  Requirement for oxygen therapy and the highest level of escalation within the first 60 minutes after extubation, including nasal cannula, simple face mask, reservoir mask, or more advanced oxygen delivery devices as clinically indicated.
Incidence of postoperative nausea and vomiting | First 60 minutes after extubation
  Incidence of postoperative nausea and vomiting occurring within the first 60 minutes after extubation. Nausea and vomiting are recorded as present or absent during the assessment period.
Patient satisfaction | At 24 hours after surgery (± 2 hours)
  Patient satisfaction with anesthetic care at 24 hours after surgery, assessed using a 0-10 numerical rating scale (NRS), where 0 indicates complete dissatisfaction and 10 indicates complete satisfaction. The recorded value represents the patient's reported score at the 24-hour assessment.
Incidence of extubation-related adverse events | From arrival in the PACU until discharge from the PACU, assessed up to 6 hours after PACU arrival.
  Incidence of extubation-related adverse events during the post-anesthesia care unit (PACU) stay, including bronchospasm, laryngospasm, reintubation, and post-obstructive pulmonary edema. Events are recorded as present or absent throughout the PACU monitoring period. The PACU stay typically lasts 2-3 hours depending on discharge criteria.

OTHER OUTCOMES:
Duration of stay in the post-anesthesia care unit (PACU) | From arrival in the PACU until discharge from the PACU, assessed up to 6 hours after PACU arrival.
  Total duration of stay in the post-anesthesia care unit (PACU), recorded in minutes from arrival in PACU until discharge based on standard discharge criteria. The PACU stay typically lasts 2-3 hours depending on discharge criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Somdetphraphutthaloetla hospital, Samut Sakhon, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the ethics committee approval and institutional data governance policies do not allow external sharing of identifiable or de-identified participant-level data. Access to study data is restricted to the research team to protect participant confidentiality and comply with local regulatory requirements.

REFERENCES:
- [Result] Young CC, Harris EM, Vacchiano C, Bodnar S, Bukowy B, Elliott RRD, Migliarese J, Ragains C, Trethewey B, Woodward A, Gama de Abreu M, Girard M, Futier E, Mulier JP, Pelosi P, Sprung J. Lung-protective ventilation for the surgical patient: international expert panel-based consensus recommendations. Br J Anaesth. 2019 Dec;123(6):898-913. doi: 10.1016/j.bja.2019.08.017. Epub 2019 Oct 3. PMID 31587835
- [Result] Blackwelder WC. "Proving the null hypothesis" in clinical trials. Control Clin Trials. 1982 Dec;3(4):345-53. doi: 10.1016/0197-2456(82)90024-1. PMID 7160191
- [Result] Langeron O, Masso E, Huraux C, Guggiari M, Bianchi A, Coriat P, Riou B. Prediction of difficult mask ventilation. Anesthesiology. 2000 May;92(5):1229-36. doi: 10.1097/00000542-200005000-00009. PMID 10781266
- [Result] Farrington CP, Manning G. Test statistics and sample size formulae for comparative binomial trials with null hypothesis of non-zero risk difference or non-unity relative risk. Stat Med. 1990 Dec;9(12):1447-54. doi: 10.1002/sim.4780091208. PMID 2281232
- [Result] Tung A, Fergusson NA, Ng N, Hu V, Dormuth C, Griesdale DGE. Pharmacological methods for reducing coughing on emergence from elective surgery after general anesthesia with endotracheal intubation: protocol for a systematic review of common medications and network meta-analysis. Syst Rev. 2019 Jan 24;8(1):32. doi: 10.1186/s13643-019-0947-2. PMID 30678727
- [Result] Minogue SC, Ralph J, Lampa MJ. Laryngotracheal topicalization with lidocaine before intubation decreases the incidence of coughing on emergence from general anesthesia. Anesth Analg. 2004 Oct;99(4):1253-1257. doi: 10.1213/01.ANE.0000132779.27085.52. PMID 15385385
- [Result] L'Hermite J, Wira O, Castelli C, de La Coussaye JE, Ripart J, Cuvillon P. Tracheal extubation with suction vs. positive pressure during emergence from general anaesthesia in adults: A randomised controlled trial. Anaesth Crit Care Pain Med. 2018 Apr;37(2):147-153. doi: 10.1016/j.accpm.2017.07.005. Epub 2017 Sep 4. PMID 28882741
- [Result] Radkowski P, Oniszczuk H, Opolska J, Pawluczuk M, Samiec M, Mieszkowski M. A Review of Non-Cardiac Complications of General Anesthesia: The Current State of Knowledge. Med Sci Monit. 2025 Apr 17;31:e947561. doi: 10.12659/MSM.947561. PMID 40241288
- [Result] Hartley M, Vaughan RS. Problems associated with tracheal extubation. Br J Anaesth. 1993 Oct;71(4):561-8. doi: 10.1093/bja/71.4.561. No abstract available. PMID 8260307
- [Result] Difficult Airway Society Extubation Guidelines Group; Popat M, Mitchell V, Dravid R, Patel A, Swampillai C, Higgs A. Difficult Airway Society Guidelines for the management of tracheal extubation. Anaesthesia. 2012 Mar;67(3):318-40. doi: 10.1111/j.1365-2044.2012.07075.x. PMID 22321104
- [Result] Benham-Hermetz J, Mitchell V. Safe tracheal extubation after general anaesthesia. BJA Educ. 2021 Dec;21(12):446-454. doi: 10.1016/j.bjae.2021.07.003. Epub 2021 Aug 25. No abstract available. PMID 34840816
- [Result] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488